CLINICAL TRIAL: NCT06886009
Title: A Regulatory Requirement Non-interventional Study to Monitor the Safety and Effectiveness of Spesolimab in Korean Patients With Flares With Generalized Pustular Psoriasis
Brief Title: Spesolimab Post-marketing Surveillance in Korean Patients With Flares With Generalized Pustular Psoriasis
Status: Not yet recruiting | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1368-0122
Record Dates: First submitted 2025-03-19; First posted 2025-03-20 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Generalized Pustular Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — spesolimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with flares with generalized pustular psoriasis (GPP)
  Interventions: Drug: Spevigo®

INTERVENTIONS:
Drug: Spevigo® — Intravenous
  Other Names: Spesolimab

SUMMARY:
The primary and secondary objectives are to respectively monitor the safety and effectiveness of Spesolimab IV in Korean patients with flares with generalized pustular psoriasis (GPP) in a routine medical practice.

ELIGIBILITY:
Inclusion criteria:

* Patients starting Spesolimab IV for the first time in accordance with the approved label in Korea (complete enumeration for the first 2 years after product launch)
* Patients with generalized pustular psoriasis (GPP) flare
* Age >/=19 years at enrolment
* Patients who have signed the data release consent form

Exclusion criteria:

* Patients with Severe or life-threatening hypersensitivity to Spesolimab or to any of the excipients
* Patients with clinically important active infections (e.g. active tuberculosis)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with generalized pustular psoriasis (GPP) in Korea
Sampling Method: Non-Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2026-02-27 (Estimated); Primary Completion 2029-06-08 (Estimated); Study Completion 2029-06-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 24 weeks
Incidence of adverse drug reactions (ADRs) | Up to 24 weeks
Incidence of serious adverse events (SAEs) | Up to 24 weeks
Incidence of serious adverse drug reactions (SADRs) | Up to 24 weeks
Incidence of unexpected adverse drug reactions | Up to 24 weeks
Incidence of adverse events of special interest (AESIs) | Up to 24 weeks
Incidence of adverse events leading to temporary or permanent discontinuation | Up to 24 weeks
Incidence of adverse events leading to death | Up to 24 weeks

SECONDARY OUTCOMES:
Physician's Global Assessment for Generalized Pustular Psoriasis (GPPGA) pustulation sub-score of 0 indicating no visible pustules at Week 1 | At Week 1
  The GPPGA is a modified the Physician's Global Assessment (PGA), a physician's assessment of psoriatic lesions, which was adapted to the evaluation of Generalized Pustular Psoriasis (GPP) patients. The investigator scores the erythema, pustules, and scaling of all GPP lesions from 0 to 4. Each component is graded separately, the average is calculated, and the final GPPA is determined from this composite score. A lower score indicates a lesser severity, with 0 being clear and 1 being almost clear.
A GPPGA pustulation sub-score of 0 indicating no visible pustules at Week 4 | At Week 4
  The GPPGA is a modified the Physician's Global Assessment (PGA), a physician's assessment of psoriatic lesions, which was adapted to the evaluation of Generalized Pustular Psoriasis (GPP) patients. The investigator scores the erythema, pustules, and scaling of all GPP lesions from 0 to 4. Each component is graded separately, the average is calculated, and the final GPPA is determined from this composite score. A lower score indicates a lesser severity, with 0 being clear and 1 being almost clear.
A GPPGA score of 0 or 1 at Week 1 | At Week 1
  The GPPGA is a modified the Physician's Global Assessment (PGA), a physician's assessment of psoriatic lesions, which was adapted to the evaluation of Generalized Pustular Psoriasis (GPP) patients. The investigator scores the erythema, pustules, and scaling of all GPP lesions from 0 to 4. Each component is graded separately, the average is calculated, and the final GPPA is determined from this composite score. A lower score indicates a lesser severity, with 0 being clear and 1 being almost clear.
A GPPGA score of 0 or 1 at Week 4 | At Week 4
  The GPPGA is a modified the Physician's Global Assessment (PGA), a physician's assessment of psoriatic lesions, which was adapted to the evaluation of Generalized Pustular Psoriasis (GPP) patients. The investigator scores the erythema, pustules, and scaling of all GPP lesions from 0 to 4. Each component is graded separately, the average is calculated, and the final GPPA is determined from this composite score. A lower score indicates a lesser severity, with 0 being clear and 1 being almost clear.

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - Pusan National University Yangsan Hospital, Busan
  - Ajou University Hospital, Gyeonggi-do
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com